CLINICAL TRIAL: NCT03260348
Title: Epidemiology and Long-term Outcomes of Patients With Acute Respiratory Distress Syndrome in Taiwan
Brief Title: Acute Respiratory Distress Syndrome in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701188B0
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study enrolls ARDS patients in medical ICUs in 11 Hospitals in Taiwan. The epidemiology and long-term outcomes of the patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients in medical intensive care unit in Sep., 2017 and Jan., 2018.

Exclusion Criteria:

* Age less than 18 years.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in medical intensive care unit during study period.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiology | two months
  The incidence of ARDS in intensive care unit
Mortality | 90 days
  The mortality rate of patients in hospital
Long-term outcome | 5 years
  Performance status of live patients discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chin Kao, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No